CLINICAL TRIAL: NCT01539616
Title: A Multicentric Prospective Randomized Double Blind Parallel Group Active Controlled Study to Evaluate the Safety and Efficacy of ZYH7 Compared to Fenofibrate in Patients With Dyslipidemia
Brief Title: A Clinical Trial to Evaluate the Safety and Efficacy of ZYH7 Compared to Fenofibrate in Patients With Dyslipidemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zydus Lifesciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZYH7.10.001.01; CTRI/2011/11/002147 (Registry Identifier: Clinical Trials Registry - India)
Record Dates: First submitted 2012-02-22; First posted 2012-02-27 (Estimated); Last update posted 2013-10-28 (Estimated); Status verified 2013-10

CONDITIONS: Hypertriglyceridemia; Dyslipidemia
Keywords: Hypertriglyceridemia; Dyslipidemia
MeSH Terms: conditions — Hypertriglyceridemia; Dyslipidemias | interventions — Fenofibrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ZYH7 4mg (Experimental): ZYH7 4mg
  Interventions: Drug: ZYH7
- ZYH7 8mg (Experimental): ZYH7 8mg
  Interventions: Drug: ZYH7
- ZYH7 16mg (Experimental): ZYH7 16mg
  Interventions: Drug: ZYH7
- Fenofibrate 160mg (Active Comparator): Fenofibrate 160mg
  Interventions: Drug: Fenofibrate

INTERVENTIONS:
Drug: ZYH7 — ZYH7 4mg given once orally in the morning before breakfast, for 8 weeks.
  Arms: ZYH7 4mg
Drug: ZYH7 — ZYH7 8 mg given once orally in the morning before breakfast, for 8 weeks.
  Arms: ZYH7 8mg
Drug: ZYH7 — ZYH7 16 mg given once orally in the morning before breakfast, for 8 weeks.
  Arms: ZYH7 16mg
Drug: Fenofibrate — Fenofibrate 160 mg given once orally in the morning before breakfast, for 8 weeks.
  Arms: Fenofibrate 160mg

SUMMARY:
ZYH7, a novel peroxisome proliferator-activated receptor (PPAR) alpha agonist, is expected to decrease triglyceride level and also correct dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years
2. Subjects of either gender, males or females
3. Triglycerides between 200 to 500 mg/dl on screening visit.
4. Body mass index (BMI) > 23 kg/m2
5. If subject is diabetic, he should be controlled on a maximum of two oral anti diabetic agents except Thiazolidinedione.
6. Subject has given informed consent for participation in this trial.

Exclusion Criteria:

1. Pregnancy and lactation.
2. History of 5% weight loss in past 6 months.
3. Subjects on treatment with insulin and PPAR alpha or gamma agonist in the past 3 month.
4. Subjects having unstable angina, acute myocardial infarction in past 3 months or heart failure of New York Heart Association (NYHA) class (III-IV).
5. Uncontrolled hypertension (150/100 mm of Hg).(If Subject using Thiazides, ACE inhibitors, beta blockers they should be on minimum 3 month stable therapy and treatment not expected to change during trial participation)
6. History of clinically significant edema.
7. History of pancreatitis or gall stone diseases.
8. Subject having thyroid-stimulating hormone (TSH) levels outside normal reference range, Subjects who are clinically euthyroid and on stable thyroid replacement therapy for 2 months prior to screening and who are anticipated to remain on this dose throughout the trial period will be allowed.
9. Uncontrolled diabetes (HbA1c ≥ 9 gm %).
10. History of active liver disease or hepatic dysfunction demonstrated by aspartate aminotransferase (AST) and Alanine Aminotransferase(ALT) ≥ 2.5 times of upper normal limit (UNL) or bilirubin ≥ 2 times UNL in the past 3 months.
11. Renal dysfunction demonstrated by abnormal Glomerular Filtration Rate (GFR) (60 ml/min) or presence of ketonuria.
12. History of myopathies or evidence of active muscle diseases demonstrated by Creatinine Phosphokinase(CPK) ≥ 10 times UNL.
13. History of any other concurrent serious illness (e.g. tuberculosis, Human Immunodeficiency Virus(HIV) infection, malignancy, etc).
14. History of alcohol and/or drug abuse.
15. History of known allergy, sensitivity or intolerance to the study drugs and their formulation ingredients.
16. Subjects on any other lipid lowering medications. (Appendix I).
17. If on contraceptive or hormone replacement therapy (HRT), therapy started or changed in last 3 months.
18. Prolonged use of steroids (15 days) in last 3 months (topical preparations, nasal and intra-articular administration are permitted).
19. History of long term use of non-steroidal anti-inflammatory drugs. (1 month)
20. Participation in any other clinical trial in the past 3 months
21. Unable to give informed consent and follow protocol requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2011-11; Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Percentage change in mean triglyceride level from baseline | 4 and 8 weeks
  Percentage change in mean triglyceride levels from baseline within and across each treatment of ZYH7 The changes will be compared with fenofibrate 160mg.

SECONDARY OUTCOMES:
Percentage change from baseline in lipid parameters | 4 and 8 weeks
  Percentage change from baseline in the following lipid parameters:
  1. Low Density Lipoprotein Cholesterol(LDL)
  2. Very Low Density Lipoprotein Cholesterol (VLDL)
  3. High Density Lipoprotein (HDL)
  4. Total cholesterol
  5. Non HDL Cholesterol (Measured value)
  6. Apo A
  7. Apo B
  8. High sensitive C-Reactive Protein (hs-CRP)

CONTACTS AND LOCATIONS:
Overall Officials: Rajendra H Jani, Ph.D (Medical), Study Director — Head & Senior Vice President, Clinical R&D, Cadila Healthcare Limited
Locations (18):
- India (18):
  - Vijayratna Diabetes Diagnosis & Treatment Centre, Upper Ground Floor, Sumeru Centre, Nr Parimal Underbridge, Paldi, Ahmedabad, Gujarat
  - Devi Hospital,Ground floor, Naranpura, Ahmedabad, Gujarat
  - Private clinic, 4, Stadium House, Ground Floor, Navrangpura, Ahmedabad, Gujarat
  - Dia Care Reseach, 1&2- Gandhi Park Society, Nr. Nehrunagar Cross Roads, Ambawadi, Ahmedabad, Gujarat
  - Govt. Medical College, Bhavnagar, Bhavnagar, Gujarat
  - Gastrocare Clinic,Ground floor, Karansinhji Main Road,, Rajkot, Gujarat
  - Balaji Hospital,First floor,clinical research department, Opp. Vidya Vikas School, Subhanpura,, Vadodara, Gujarat
  - Pace Clinical Research (A. Unit of Pranav Diabetes Centre), No. 53, Nanda Complex, Ramamurthy Nagar Main Road, Banasawadi, Bangalore, Karnataka
  - Srinivasa clinic and Diabetic Care centre, 197, 2nd floor, Near Avalahalli BDA park, BSK 3rd stage, Bangalore, Karnataka
  - Mallige Healthcare Centre, # 402, 8th main, 8th cross, Near Dr. M. C. Modi Compound. P.J.EXTN,, Davangere, Karnataka
  - Deogiri Diabetes Centre, 46 Samata Nagar, Near Kranti Chowk Police Station, Aurangabad, Maharashtra
  - Bhatia Hospital, Tardeo Road,Room no 19, Basement floor,Research room,, Mumbai, Maharashtra
  - Pai Clinic & Diagnostic Centre - Abhinav Apartments, 778/B-4, First floor, Shivajinagar, Next to Congress House, Pune, Maharashtra
  - Shree Nidan Hospital, Clinical trial department, First floor, 27-28 Vidhyut nagar-A, Ajmer road, Jaipur, Rajasthan
  - Aruna Diabetes Centre, 56,Thiruvengatapuram, Near Nungambakkam Railway Station, Choolamedu, Chennai, Tamil Nadu
  - Mother's Care Diabetes Centre, Room no 9, Phase 1, Sathuvachari, Vellore, Tamil Nadu
  - Department of Endocrinology, Room No.9, 4 th Floor, Ronald Ross Building, Institute of Post Graduate Medical Education & Research, 244 AJC Bose Road., Kolkata, West Bengal
  - Room no 3027,Research block B,Department of Endocrinology PGIMER, Chandigarh